CLINICAL TRIAL: NCT00622843
Title: An Open-Label, Phase III, Randomized Study of Pneumococcal Conjugate Vaccination in HIV, in Comparison to Polysaccharide Vaccine Boosting in Previously Vaccinated Patients
Brief Title: Pneumococcal Conjugate Vaccination in HIV in Comparison to Polysaccharide Vaccine Boosting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); US Military HIV Research Program (Network); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Agan, Deputy Science Director, IDCRP, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RV150 Prevnar
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Streptococcus Pneumoniae
Keywords: pneumococcal conjugate vaccine; polysaccharide vaccine; PPV; PCV; Streptococcus pneumoniae; Prevnar; Pneumovax; HIV
MeSH Terms: conditions — HIV Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): PCV, 210 patients
  Interventions: Biological: pneumococcal conjugate vaccine
- Group 2 (Active Comparator): PPV, 110 patients
  Interventions: Biological: pneumococcal polysaccharide vaccine
- Group 3 (Active Comparator): PCV, HIV-negative, 25 patients
  Interventions: Biological: pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: pneumococcal conjugate vaccine — Prevnar is manufactured as a liquid preparation. Each 0.5 mL dose is formulated to contain:
  2 μg of each saccharide for serotypes 4, 9V, 14, 18C, 19F, and 23F, and 4 μg of serotype 6B per dose (16 μg total saccharide); approximately 20 μg of CRM197 carrier protein; and 0.125 mg of aluminum per 0.5 mL dose as aluminum phosphate adjuvant. After shaking, the vaccine is a homogeneous, white suspension.
  Other Names: PCV
  Arms: Group 1; Group 3
Biological: pneumococcal polysaccharide vaccine — PNEUMOVAX 23 is manufactured according to methods developed by the Merck Research Laboratories. Each 0.5 mL dose of vaccine contains 25 μg of each polysaccharide type in isotonic saline solution containing 0.25% phenol as a preservative.
  Other Names: PPV
  Arms: Group 2

SUMMARY:
Purpose: To study the immune response of the newly licensed pneumococcal conjugate vaccine (PCV) in comparison to the pneumococcal polysaccharide vaccine (PPV) to determine if a significantly better immunologic response to boosting can be elicited in patients previously vaccinated with PPV.

ELIGIBILITY:
Inclusion Criteria for HIV positive subjects:

1. At least one prior PPV ≥ 3 and < 8 years ago, while HIV positive. There is no upper limit to the number of previously received PPVs.
2. HIV-positive (except 25 HIV-negative persons as control group).
3. Age between 18 and 60 years of age.
4. Availability of patient to remain within the immediate area for the period of the study and be able to comply with protocol requirements.

Exclusion Criteria for HIV positive subjects:

1. Prior allergic reaction to the PPV
2. Allergic to components of PCV, including diphtheria toxin.
3. Pregnant or lactating females as defined by history or positive HCG urine test.
4. History of chronic viral hepatitis or biochemical evidence to include pretreatment AST or ALT values greater than 3 fold higher than upper limit of normal, or a creatinine of greater than 1.8 mg/dl
5. History of splenectomy
6. Temperature of >38C
7. Inability to ambulate for more than 1000 meters secondary to fatigue, pain or weakness.
8. Patients in whom IM vaccination is not possible because of disease or medication. (e.g. hemophilia, coumadin therapy).
9. Patients diagnosed with HIV wasting disease
10. Viral load over 50,000 copies/ml.
11. History or evidence of recent illicit drug or alcohol abuse.
12. Use of immunosuppressive agents, to include corticosteroids and cancer chemotherapeutic agents.

Inclusion Criteria for HIV negative subjects:

1. HIV-negative by HIV ELISA within the last 12 months
2. Age between 18 and 60 years of age.
3. Availability of patient to remain within the immediate area for the period of the study and be able to comply with protocol requirements.

Exclusion Criteria for HIV negative subjects:

1. Prior PCV and/or PPV vaccination.
2. Prior allergic reaction to the PPV
3. Allergic to components of PCV, including diphtheria toxin.
4. Pregnant or lactating females as defined by history or positive HCG urine test.
5. History of chronic viral hepatitis or biochemical evidence to include pretreatment AST or ALT values greater than 3 fold higher than upper limit of normal, or a creatinine of greater than 1.8 mg/dl
6. History of splenectomy
7. Temperature of >38C
8. Inability to ambulate for more than 1000 meters secondary to fatigue, pain or weakness.
9. Patients in whom IM vaccination is not possible because of disease or medication. (e.g. hemophilia, coumadin therapy).
10. History or evidence of recent illicit drug or alcohol abuse.
11. Use of immunosuppressive agents, to include corticosteroids and cancer chemotherapeutic agents.
12. Works in chain of command of primary/associate investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2002-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Agan, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (6):
- United States (6):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Tripler Army Medical Center, Tripler AMC, Hawaii
  - National Naval Medical Center, Bethesda, Maryland
  - San Antonio Military Medical Center, Lackland Air Force Base, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

REFERENCES:
- [Result] Crum-Cianflone NF, Roediger M, Huppler Hullsiek K, Ganesan A, Landrum M, Weintrob A, Agan B, Medina S, Rahkola J, Hale B, Janoff EN; Infectious Disease Clinical Research Program HIV Working Group. The association of ethnicity with antibody responses to pneumococcal vaccination among adults with HIV infection. Vaccine. 2010 Nov 10;28(48):7583-8. doi: 10.1016/j.vaccine.2010.09.056. Epub 2010 Sep 29. PMID 20887830
- [Result] Crum-Cianflone NF, Huppler Hullsiek K, Roediger M, Ganesan A, Patel S, Landrum ML, Weintrob A, Agan BK, Medina S, Rahkola J, Hale BR, Janoff EN; Infectious Disease Clinical Research Program HIV Working Group. A randomized clinical trial comparing revaccination with pneumococcal conjugate vaccine to polysaccharide vaccine among HIV-infected adults. J Infect Dis. 2010 Oct 1;202(7):1114-25. doi: 10.1086/656147. PMID 20795819

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 345 is the number of potential subjects that was approved for enrollment by the IRB (Group 1 PCV = 210; Group 2 PPV = 110; Group 3 HIV-negative = 25). 275 is the total number of subjects who actually consented to participate. 229 is the number of subject who were vaccinated. In 2008, the DSMB voted unanimously to recommend no further enrollment.
Groups:
- Group 1 - PCV: PCV, 210 patients
  pneumococcal conjugate vaccine: Prevnar is manufactured as a liquid preparation. Each 0.5 mL dose is formulated to contain: 2 μg of each saccharide for serotypes 4, 9V, 14, 18C, 19F, and 23F, and 4 μg of serotype 6B per dose (16 μg total saccharide); approximately 20 μg of CRM197 carrier protein; and 0.125 mg of aluminum per 0.5 mL dose as aluminum phosphate adjuvant. After shaking, the vaccine is a homogeneous, white suspension.
- Group 2 - PPV: PPV, 110 patients
  pneumococcal polysaccharide vaccine: PNEUMOVAX 23 is manufactured according to methods developed by the Merck Research Laboratories. Each 0.5 mL dose of vaccine contains 25 μg of each polysaccharide type in isotonic saline solution containing 0.25% phenol as a preservative.
- Group 3 - HIV-negative: PCV, HIV-negative, 25 patients
  pneumococcal conjugate vaccine: Prevnar is manufactured as a liquid preparation. Each 0.5 mL dose is formulated to contain: 2 μg of each saccharide for serotypes 4, 9V, 14, 18C, 19F, and 23F, and 4 μg of serotype 6B per dose (16 μg total saccharide); approximately 20 μg of CRM197 carrier protein; and 0.125 mg of aluminum per 0.5 mL dose as aluminum phosphate adjuvant. After shaking, the vaccine is a homogeneous, white suspension.
Period: Overall Study
Arm/Group | Group 1 - PCV | Group 2 - PPV | Group 3 - HIV-negative
Started | 131 | 73 | 25
Completed | 131 | 73 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 131 | 73 | 25 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 131 | 73 | 25 | 229
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 7 | 21
  Male | 120 | 70 | 18 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 3 | 26
  Not Hispanic or Latino | 119 | 62 | 22 | 203
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 50 | 27 | 2 | 79
  White | 71 | 40 | 21 | 132
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 131 | 73 | 25 | 229
CDC stage [Count of Participants; unit: Participants] — Centers for Disease Control and Prevention (CDC) stage of human immunodeficiency virus (HIV) infection. HIV infection stage, based on age-specific CD4+ T-lymphocyte count or CD4+ T-lymphocyte percentage of total lymphocytes.
  6 years through adult: A = asymptomatic, acute (primary) HIV or persistent generalized lymphadenopathy (PGL), ≥500 cells/µL (≥26%); B = symptomatic, not (A) or (C) conditions, 200-499 cells/µL (14-25%); C = acquired immunodeficiency syndrome (AIDS) indicator conditions, <200 cells/µL (<14%) Population: CDC stage only applies to the HIV-infected arms of the study. This baseline measure is not applicable to the HIV-negative arm.
  Participants
    number analyzed (Participants) | 131 | 73 | 0 | 204
    A | 91 | 55 |  | 146
    B | 25 | 9 |  | 34
    C | 15 | 9 |  | 24
CD4 T cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: CD4 T cell count only applies to the HIV-infected arms of the study. This baseline measure is not applicable to the HIV-negative arm.
  cells/mm^3
    number analyzed (Participants) | 131 | 73 | 0 | 204
    (all) | 533 [396 to 700] | 513 [388 to 714] |  | 533 [391 to 701]
Current receipt of HAART [Count of Participants; unit: Participants] — Highly active antiretroviral therapy (HAART) Population: HAART only applies to the HIV-infected arms of the study. This baseline measure is not applicable to the HIV-negative arm.
  Participants
    number analyzed (Participants) | 131 | 73 | 0 | 204
    (all) | 111 | 56 |  | 167
IgG levels at baseline [Median (Inter-Quartile Range); unit: ng/mL] — For the Total column, the medians and IQRs reported are weighted averages of the median, IQR1, and IQR3 from the three groups.
  ng/mL
    Serotype 4 | 293 [108 to 793] | 254 [105 to 580] | 264 [108 to 595] | 277 [107 to 703]
    Serotype 9V | 556 [258 to 1389] | 425 [237 to 1269] | 746 [488 to 1437] | 535 [276 to 1356]
    Serotype 14 | 860 [321 to 5039] | 771 [218 to 3083] | 254 [99 to 564] | 765 [264 to 3927]
    Serotype 19F | 723 [329 to 1971] | 480 [239 to 1154] | 737 [182 to 1127] | 647 [284 to 1618]

OUTCOME MEASURES:

1. Primary Outcome: Positive Immune Responses in the Human Immunodeficiency Virus (HIV)-Infected Pneumococcal Conjugate Vaccine (PCV) and Pneumococcal Polysaccharide Vaccine (PPV) Arms
Description: The primary end point is greater than or equal to a 2-fold increase in the IgG level for at least 2 of the 4 serotypes on day 60, with levels greater than or equal to 1000 ng/mL.
Time Frame: Day 14, 60, and 180 after vaccination
Population: The number of participants analyzed represents the number of participants who were actually vaccinated from those who consented to participate.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PCV | Group 2 - PPV | Group 3 - HIV-negative
Number analyzed (Participants) | 131 | 73 | 25
Participants
  Day 14 : At least 2 of 4 serotypes | 67 | 23 | 22
  Day 14 : At least 3 of 4 serotypes | 37 | 11 | 16
  Day 14 : Serotype 4 | 54 | 17 | 17
  Day 14 : Serotype 9V | 68 | 22 | 22
  Day 14 : Serotype 14 | 57 | 27 | 18
  Day 14 : Serotype 419F | 37 | 12 | 14
  Day 60 : At least 2 of 4 serotypes | 68 | 23 | 22
  Day 60 : At least 3 of 4 serotypes | 37 | 9 | 16
  Day 60 : Serotype 4 | 48 | 15 | 18
  Day 60 : Serotype 9V | 63 | 25 | 21
  Day 60 : Serotype 14 | 61 | 28 | 18
  Day 60 : Serotype 419F | 42 | 12 | 20
  Day 180 : At least 2 of 4 serotypes | 47 | 30 | 21
  Day 180 : At least 3 of 4 serotypes | 26 | 11 | 16
  Day 180 : Serotype 4 | 37 | 16 | 18
  Day 180 : Serotype 9V | 49 | 24 | 22
  Day 180 : Serotype 14 | 47 | 22 | 18
  Day 180 : Serotype 419F | 38 | 13 | 12

2. Primary Outcome: Adverse Events (AEs) Occurring Temporally (Within 7 Days) in Association With Pneumococcal Vaccination
Time Frame: Day 7 after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PCV | Group 2 - PPV | Group 3 - HIV-negative
Number analyzed (Participants) | 131 | 73 | 25
Participants
  Number of AEs = 0 | 80 | 50 | 1
  Number of AEs =1 | 36 | 17 | 13
  Number of AEs >/= 2 | 15 | 6 | 11

3. Secondary Outcome: Assessment of CD4+ Cell Count Changes Caused by Vaccination With PCV and PPV.
Description: The pairwise change in CD4+ cell count from the time of screening to each time frame (day 14, day 60 and day 180 post-vaccination) (CD4+ cell count at day 14/60/180 [minus] CD4+ cell count at screening).
  Analysis Population Description (further details): not all participants completed each follow-up visit. Therefore, a different number of participants analyzed is noted for each visit day. For example, in Group 1, 131 participants completed the screening visit but only 129 completed Day 14, and only 123 completed Day 60, etc.
Time Frame: Day 14, 60, and 180 after vaccination
Population: Number of participants analyzed for each time frame: Group 1 (Day 14=129/131; Day 60=123/131; Day 180=119/131); Group 2 (Day 14=69/73; Day 60=67/73; Day 180=67/73). Group 3 = 0 since these data are not applicable to HIV-negative subjects.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 131 | 73 | 0
cells/mm^3
  Day 14 (CD4): number analyzed (Participants) | 129 | 69 | 0
  Day 14 (CD4) | 40.17 (22.29) | 14.66 (28.08) |
  Day 60 (CD4): number analyzed (Participants) | 123 | 67 | 0
  Day 60 (CD4) | 13.20 (21.13) | 22.57 (30.73) |
  Day 180 (CD4): number analyzed (Participants) | 119 | 67 | 0
  Day 180 (CD4) | 29.65 (21.57) | 12.22 (27.81) |

4. Secondary Outcome: Assessment of the Importance of the Host Immune Status (CD4+ Count) on the PCV and PPV Immunologic Response.
Description: Number with ≥ Successes, which is defined as: Success = 2-fold increase on Log10 scale -- if log10(Day 60) - log10(Screening) > log10(2)
Time Frame: Day 60 after vaccination
Population: The number analyzed in the rows is based on the number of participants who had the CD4+ counts in each category at baseline. This data is not applicable to Group 3 since they are HIV-negative.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - PCV | Group 2 - PPV | Group 3 - HIV-negative
Number analyzed (Participants) | 131 | 73 | 0
Participants
  </= 350 cells/mm^3: number analyzed (Participants) | 21 | 9 | 0
  </= 350 cells/mm^3 | 8 | 5 |
  351-500 cells/mm^3: number analyzed (Participants) | 35 | 26 | 0
  351-500 cells/mm^3 | 22 | 13 |
  501-750 cells/mm^3: number analyzed (Participants) | 53 | 24 | 0
  501-750 cells/mm^3 | 38 | 12 |
  >/= 751 cells/mm^3: number analyzed (Participants) | 22 | 14 | 0
  >/= 751 cells/mm^3 | 14 | 5 |

5. Secondary Outcome: Assessment of Viral Load Changes Caused by Vaccination With PCV and PPV.
Description: The pairwise change in viral load from the time of screening to each time frame (day 14, day 60 and day 180 post-vaccination), similar to CD4 change above.
Time Frame: Day 14, 60, and 180 after vaccination
Population: Number of participants analyzed for each time frame: Group 1 (Day 14=129/131; Day 60=123/131; Day 180=117/131); Group 2 (Day 14=70/72; Day 60=68/72; Day 180=68/72). Group 3 = 0 since these data are not applicable to HIV-negative subjects.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 131 | 72 | 0
log10 copies/mL
  Day 14 (viral load): number analyzed (Participants) | 129 | 70 | 0
  Day 14 (viral load) | -0.02 (0.08) | 0.03 (0.12) |
  Day 60 (viral load): number analyzed (Participants) | 123 | 68 | 0
  Day 60 (viral load) | -0.05 (0.08) | 0.08 (0.14) |
  Day 180 (viral load): number analyzed (Participants) | 117 | 68 | 0
  Day 180 (viral load) | -0.03 (0.09) | 0.01 (0.13) |

ADVERSE EVENTS:
Time Frame: Baseline to 180 days post vaccination.
Arm/Group | Group 1 - PCV | Group 2 - PPV | Group 3 - HIV-negative
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/73 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/73 | 0/25
Other Adverse Events (participants affected / at risk) | 51/131 | 23/73 | 24/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - PCV (N=131) | Group 2 - PPV (N=73) | Group 3 - HIV-negative (N=25)
Local tenderness (Musculoskeletal and connective tissue disorders) | 36 | 14 | 23
Malaise (General disorders) | 5 | 3 | 7
Myalgia (General disorders) | 11 | 7 | 5
Headache (General disorders) | 3 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Local swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Local site reaction (Skin and subcutaneous tissue disorders) | 7 | 1 | 3
Injection site, other (General disorders) | 3 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Dizziness (General disorders) | 0 | 3 | 0
Other related (General disorders) | 1 | 1 | 3

LIMITATIONS AND CAVEATS:
Limitations include: enrollment halted before full recruitment, no defined correlate of protective pneumococcal immunity in adults, prior pneumococcal vaccination may result in blunted responses to subsequent vaccination, and limiting to 4 serotypes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No